CLINICAL TRIAL: NCT01630603
Title: Maternal Vitamin D Status and Neonatal Bone Strength
Acronym: Vitamin D
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MMC14-12
Record Dates: First submitted 2012-06-18; First posted 2012-06-28 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2012-06

CONDITIONS: Maternal Vitamin D Status; Neonatal Bone Quantitative Ultrasound Measurements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- mother infants pairs

SUMMARY:
Objectives:

1. To determine the incidence of vitamin D deficiency among Israeli pregnant women
2. To access whether maternal vitamin D status affects infant bone strength.

Methods:

1. Vitamin D levels -in cord blood and maternal blood
2. The mother will fill a demographic and nutritional questionnaire

   The Infants:
3. Growth assessment of the infants: weight length and head circumference
4. Bone strength measurement by Quantitative Ultrasound (Sunlight Omnisense 7000/8000TM)

ELIGIBILITY:
Inclusion Criteria:

* mother-baby pairs,
* birth week 35-42.
* Jewish and Arab women that read and understand Hebrew.

Exclusion Criteria:

* large neonatal congenital defects.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inborn mother infants pairs
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-07; Primary Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Bone speed of sound and maternal vitamin D levels | first tow days of life

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Meir Medical Center, Kfar Saba
  - Neonatal department Meir Medical Center, Kfar Saba